CLINICAL TRIAL: NCT02660801
Title: Spinal Manipulation and Spinal Mobilization Effects in Participants With and Without Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Fonds de la Recherche en Santé du Québec (Other Government); Unité de recherche en santé musculosqulettique (Unknown)
Responsible Party: Principal Investigator, Martin Descarreaux, Dr Martin Descarreaux DC, PhD, Université du Québec à Trois-Rivières
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UQTR-2016-STIF
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Back Pain
Keywords: spinal manipulation; spinal mobilization; spinal stiffness
MeSH Terms: conditions — Back Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal manipulation (Experimental): Twenty-six participants with chronic nonspecific back pain will participate in two experimental sessions. During the first session, each participant will received either a spinal manipulation of a spinal mobilization of their thoracic spine preceded and followed by the assessment of their thoracic spine stiffness. The second session (24 to 48h after) will be identical but with the other experimental condition (spinal manipulation or spinal mobilization).
  Interventions: Procedure: Spinal manipulation
- Spinal mobilization (Experimental): Twenty-six participants with chronic nonspecific back pain will participate in two experimental sessions. During the first session, each participant will received either a spinal manipulation of a spinal mobilization of their thoracic spine preceded and followed by the assessment of their thoracic spine stiffness. The second session (24 to 48h after) will be identical but with the other experimental condition (spinal manipulation or spinal mobilization).
  Interventions: Procedure: Spinal mobilization

INTERVENTIONS:
Procedure: Spinal manipulation — A high-velocity and low-amplitude thrust delivered posteroanteriorly to a thoracic vertebra
  Other Names: SMa
  Arms: Spinal manipulation
Procedure: Spinal mobilization — Three repetitions of a low-velocity and low-amplitude nonthrust movement delivered posteroanteriorly to a thoracic vertebra
  Other Names: SMo
  Arms: Spinal mobilization

SUMMARY:
The objective of the present study is to compare the neuromechanical responses to spinal manipulation and spinal mobilization in participants with chronic nonspecific middle back pain.

DETAILED DESCRIPTION:
Although evidences suggest a similar effectiveness of spinal manipulation and spinal mobilization, there is no study that compares the neuromechanical effects of these manual therapies in a experimental context and with the standardization of both interventions. Therefore, the objective of the present study is to compare the neuromechanical responses to spinal manipulation (low-amplitude and high-velocity dynamic thrust) and spinal mobilization (repetitions of a low-amplitude and low-velocity nonthrust movement) in participants with and without chronic nonspecific back pain.

ELIGIBILITY:
Inclusion Criteria:

* presenting or not a history of chronic nonspecific back pain

Exclusion Criteria:

* History of back trauma or surgery
* Severe osteoarthritis
* Inflammatory arthritis
* Vascular conditions
* Contraindication to the use of spinal manipulation or spinal mobilization
* Pregnancy
* Scoliosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: the participants were recruited among the local community
Groups:
- Spinal Manipulation Then Spinal Mobilization: Participants first received spinal manipulation*. After a washout period of 48h, they then received a spinal mobilization* at the same spinal level.
  *Spinal manipulation is characterized by a preload force of 70 N for 500 ms leading to a peak force of 260 N in 125 ms (rate of force application: 1520 N/s) and spinal mobilization use 3 oscillatory cycles of 85 N in 800 ms (rate of force application: 106 N/s)
- Spinal Mobilization Then Spinal Manipulation: Participants first received spinal mobilization*. After a washout period of 48h, they then received a spinal manipulation* at the same spinal level.
  *Spinal manipulation is characterized by a preload force of 70 N for 500 ms leading to a peak force of 260 N in 125 ms (rate of force application: 1520 N/s) and spinal mobilization use 3 oscillatory cycles of 85 N in 800 ms (rate of force application: 106 N/s)
Period: Overall Study
Arm/Group | Spinal Manipulation Then Spinal Mobilization | Spinal Mobilization Then Spinal Manipulation
Started | 11 | 15
Completed | 11 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Experimental group 1: spinal manipulation, spinal mobilization Participants first received spinal manipulation. After a washout period of 48h, they then received a spinal mobilization at the same spinal level.
  Experimental group 2: spinal mobilization, spinal manipulation Participants first received spinal mobilization. After a washout period of 48h, they then received a spinal manipulation at the same spinal level.
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 26
Global spinal stiffness [Mean (Standard Deviation); unit: N/mm] — Spinal stiffness is the relationship between spinal displacement and the resistive force to that movement Global stiffness was defined as the slope of the straight-line best fitting the force-displacement data between 10 and 45 N
  N/mm
    Spinal Manipulation | 7.7 (1.4)
    Spinal mobilization | 7.6 (1.8)
Terminal spinal stiffness [Mean (Standard Deviation); unit: N/mm] — terminal stiffness was defined as the ratio of the variation of force and displacement between 10 and 45 N
  N/mm
    Spinal manipulation | 7.9 (1.5)
    Spinal mobilization | 7.8 (1.9)
Pressure provoked pain [Mean (Standard Deviation); unit: units on a scale] — Pressure provoked pain intensity was assessed immediately after each spinal stiffness assessment using a 0 to 100 visual analog pain scale.
  0 is no pain and 100 represents the maximum
  units on a scale
    Spinal manipulation | 47.9 (22.8)
    Spinal mobilization | 47.2 (23.2)

OUTCOME MEASURES:

1. Primary Outcome: Global Spinal Stiffness
Description: Global stiffness was defined as the slope of the straight-line best fitting the force-displacement data between 10 and 45 N
Time Frame: two-minutes before spinal manipulation delivery up to two-minutes after
Measure: Mean (Standard Deviation); unit: N/mm
Groups:
- Spinal Manipulation: SMa characterized by a preload force of 70 N for 500 ms leading to a peak force of 260 N in 125 ms (rate of force application: 1520 N/s)
- Spinal Mobilization: SMo use 3 oscillatory cycles of 85 N in 800 ms (rate of force application: 106 N/s)
Arm/Group | Spinal Manipulation | Spinal Mobilization
Number analyzed (Participants) | 26 | 26
N/mm | 7.6 (1.8) | 7.8 (1.7)

2. Primary Outcome: Terminal Spinal Stiffness
Description: Terminal stiffness was defined as the ratio of the variation of force and displacement between 10 and 45 N
Time Frame: two-minutes before spinal mobilization delivery up to two-minutes after
Measure: Mean (Standard Deviation); unit: N/mm
Arm/Group | Spinal Manipulation | Spinal Mobilization
Number analyzed (Participants) | 26 | 26
N/mm | 7.9 (1.5) | 7.8 (1.9)

3. Primary Outcome: Pressure Provoked Pain
Description: Pressure provoked pain intensity was assessed immediately after each spinal stiffness assessment using a 0 to 100 visual analog pain scale minimum value=0, maximum value=100. 0 is no pain while 100 is the worse outcome
Time Frame: immediately after the therapeutic modality application
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Spinal Manipulation | Spinal Mobilization
Number analyzed (Participants) | 26 | 26
score on a scale | 36.6 (23.7) | 45.4 (24.3)

4. Primary Outcome: Muscular Response, Superior Level Ratio
Description: To assess the muscular response during therapeutic modalities, the resulting bipolar sEMG signals were first digitally band-pass filtered using a frequency bandwidth of 20-450 Hz (2nd order Butterworth filter). For SMa, the peak root mean square (RMS) value was computed for each electrode using a 250 ms window (125 ms before and 125 ms after the peak force). The RMS values obtained for each electrode were then normalized (nRMS) to the respective RMS value calculated during the sEMG normalization trial.
Time Frame: During the spinal manipulation and mobilization
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Spinal Manipulation | Spinal Mobilization
Number analyzed (Participants) | 26 | 26
ratio | 0.78 (0.56) | 0.16 (0.09)

5. Primary Outcome: Muscular Response, Inferior Level Ratio, Normalized RMS
Description: as for outcome 4
Time Frame: During the spinal manipulation and mobilization
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Spinal Manipulation | Spinal Mobilization
Number analyzed (Participants) | 26 | 26
ratio | 0.79 (0.60) | 0.16 (0.10)

ADVERSE EVENTS:
Time Frame: 48 hours
Groups:
- Spinal Manipulation Then Spinal Mobilization: 11 participants with chronic nonspecific middle back pain will participate in two experimental sessions. During the first session, each participant received either a spinal manipulation of their thoracic spine preceded and followed by the assessment of their thoracic spine stiffness. The second session (24 to 48h after) will be identical but with spinal mobilization.
  Spinal manipulation: A high-velocity and low-amplitude thrust delivered posteroanteriorly to a thoracic vertebra
  Spinal mobilization: Three repetitions of a low-velocity and low-amplitude nonthrust movement delivered posteroanteriorly to a thoracic vertebra
- Spinal Mobilization Then Spinal Manipulation: 11 participants with chronic nonspecific middle back pain will participate in two experimental sessions. During the first session, each participant received a spinal mobilization of their thoracic spine preceded and followed by the assessment of their thoracic spine stiffness. The second session (24 to 48h after) will be identical but with spinal manipulation .
  Spinal manipulation: A high-velocity and low-amplitude thrust delivered posteroanteriorly to a thoracic vertebra
  Spinal mobilization: Three repetitions of a low-velocity and low-amplitude nonthrust movement delivered posteroanteriorly to a thoracic vertebra
Arm/Group | Spinal Manipulation Then Spinal Mobilization | Spinal Mobilization Then Spinal Manipulation
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 0/11 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT02660801/Prot_SAP_000.pdf